CLINICAL TRIAL: NCT00743249
Title: A Three-Month Safety Study to Determine the Retention Times of Side-Arm Canalicular Stents
Brief Title: Punctal Plug Study to Determine the Safety and Retention Times of Various Lengths of Canalicular Stents in Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: C-07-23
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Healthy; Dry Eye
Keywords: Dry eye; Tear duct; Punctal plug
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canalicular stent, 10 mm (Experimental): MINI MONOKA canalicular stent (tube), 10 mm, inserted in the lower lacrimal canaliculus (tear duct) of one eye for up to 3 months
  Interventions: Device: MINI MONOKA canalicular stent, 10 mm
- Canalicular stent, 20 mm (Experimental): MINI MONOKA canalicular stent (tube), 20 mm, inserted in the lower lacrimal canaliculus (tear duct) of one eye for up to 3 months
  Interventions: Device: MINI MONOKA canalicular stent, 20 mm

INTERVENTIONS:
Device: MINI MONOKA canalicular stent, 10 mm — 40 mm hollow intubation stent composed of a silicon tube and an oval collarette head (plug), cut to 10 mm length
  Other Names: MINI MONOKA
  Arms: Canalicular stent, 10 mm
Device: MINI MONOKA canalicular stent, 20 mm — 40 mm hollow intubation stent composed of a silicon tube and an oval collarette head (plug), cut to 20 mm length
  Other Names: MINI MONOKA
  Arms: Canalicular stent, 20 mm

SUMMARY:
The purpose of this study was to determine the safety and retention times of two different lengths (10 mm and 20 mm) of the MINI MONOKA canicular stent when inserted in the eye for up to three months in subjects with or without dry eye.

DETAILED DESCRIPTION:
This study consisted of 6 visits conducted over a period of 3 months. At Visit 1 (Day 0), the canalicular stent was inserted. If the stent insertion failed, the subject was rescheduled for insertion at the Day 2 visit. If the stent insertion was not successfully completed by the end of the Day 2 visit, the subject was discontinued from the study. Any subject who had the stent inserted but lost the stent (noticed or unnoticed) after the Day 2 Visit was considered to have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent.
* With or without dry eye.
* Willing to discontinue contact lenses during the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Chronic, recurrent, or severe inflammatory eye disease.
* Ocular trauma within the past 6 months.
* Ocular hypertension or glaucoma.
* History of punctal plug/canalicular stent insertion.
* Other protocol-defined exclusion criteria may apply.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Landry, Ph.D., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from four US study centers.
Period: Overall Study
Arm/Group | Canalicular Stent, 10 mm | Canalicular Stent, 20 mm
Started | 30 | 30
Completed | 28 | 24
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 4
Not completed — Patient Decision Unrelated to Ad Event | 0 | 1
Not completed — Unsuccessful insertion of stent | 2 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized participants for whom stent insertion was successfully completed (57).
Groups:
- Total: Total of all reporting groups
Arm/Group | Canalicular Stent, 10 mm | Canalicular Stent, 20 mm | Total
Number analyzed (Participants) | 28 | 29 | 57
Age Continuous [Mean (Standard Deviation); unit: years] | 63.0 (10.5) | 62.2 (10.8) | 62.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Mean Retention Time
Description: At all study visits the investigator conducted a slit lamp examination to determine whether the canalicular stent was present.
Time Frame: From baseline (Day 0) up to Month 3
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Canalicular Stent, 10 mm | Canalicular Stent, 20 mm
Number analyzed (Participants) | 28 | 29
Days | 87.4 (16.8) | 61.9 (36.0)

2. Secondary Outcome: Percentage of Subjects Retaining the Stent at Month 3
Description: as for outcome 1
Time Frame: Month 3
Population: Intent to treat
Measure: Number; unit: Percentage of subjects
Arm/Group | Canalicular Stent, 10 mm | Canalicular Stent, 20 mm
Number analyzed (Participants) | 28 | 29
Percentage of subjects | 92.9 | 48.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (3 months, 26 days)
Description: The safety population includes all subjects randomized into the study for whom an attempt to insert a canalicular stent occurred.
Arm/Group | Canalicular Stent, 10 mm | Canalicular Stent, 20 mm
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 10/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canalicular Stent, 10 mm (N=30) | Canalicular Stent, 20 mm (N=30)
Eyelids Pruritus (Eye disorders) | 2 | 2
Foreign Body Sensation in Eyes (Eye disorders) | 2 | 3
Eyelid Irritation (Eye disorders) | 1 | 3
Eyelid Oedema (Eye disorders) | 0 | 3
Lacrimation Increased (Eye disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.